CLINICAL TRIAL: NCT02197910
Title: Association Between Consumption of Different Dosages of Bioactive Wheat Peptides and Blood Pressure (BP) Level and Other Biomarkers of Cardiovascular Disease Risk in Healthy Subjects With High-normal BP: a Double-blind, Cross-over, RCT
Brief Title: Different Dosages of Bioactive Wheat Peptides and Blood Pressure Level and CVD Risk Biomarkers in Healthy Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bologna (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Claudio Borghi, Prof., University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BACCHUS_PASTATREND_2014
Record Dates: First submitted 2014-07-19; First posted 2014-07-23 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Pre-hypertension
MeSH Terms: conditions — Prehypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- High content of wheat bioactive peptides (Active Comparator): 100 gr pasta/day, containing around 15 mg bioactive peptides (High content of wheat bioactive peptides)
  Interventions: Other: Comparisons of two kind of pasta with low or high content of wheat bioactive peptides (sequence High->Low)
- Low dose of wheat bioactive peptides (Placebo Comparator): 100 gr pasta/day, containing around 3 mg bioactive peptides
  Interventions: Other: Comparisons of two kind of pasta with low or high content of wheat bioactive peptides (sequence Low->High)

INTERVENTIONS:
Other: Comparisons of two kind of pasta with low or high content of wheat bioactive peptides (sequence Low->High)
  Arms: Low dose of wheat bioactive peptides
Other: Comparisons of two kind of pasta with low or high content of wheat bioactive peptides (sequence High->Low)
  Arms: High content of wheat bioactive peptides

SUMMARY:
In this study we will assess the effects of bioactive peptide rich wheat products on blood pressure and estimated cardiovascular disease risk. This will be a pilot, explorative, cross-over, randomized double-blind 2 groups x 2-arms controlled, clinical trial. The intervention will be based on commercially-packaged pasta, which will appear and taste the same; (i) low dose bioactive peptides vs. (ii) high dose bioactive peptides. Inclusion Criteria will be: Male and female non-diabetic adult volunteers at increased estimated CV risk (ESC/EAS SCORE) with SBP 130-139 mmHg and/or DBP 85-90 mmHg); Age included between 40 and 70 years old; Primary prevention for CVD but otherwise in good general health and have had no major illness in the previous 6-months; Volunteer providing their signed and dated informed consent form. Exclusion Criteria will be: Severe medical illness/chronic disease/gastrointestinal pathology (e.g. coeliac disease); Secondary prevention for CVD; Treatment with drugs potentially affecting BP (including antihypertensive drugs) or other related CV risk factors; Consumption of nutraceuticals, botanical extracts or other vitamin supplements; Volunteer diagnosed as being hypertensive A total of 60 participants will be recruited and following adherence to a standardized diet for a 4-week period, will be randomly assigned to complete one of 2 treatment sequences by consuming a prescribed quantity of pasta products for a 4-week period followed by a 4-week washout before random assignment to the 2nd treatment.

The Primary Outcome will be the modification of office blood pressure (assessed by systolic and diastolic BP, pulse and mean pressure (mean of 3 standing & sitting measures) and 24-hour blood pressure.

Additional outcomes include: Anthropometric parameters (Weight, WC, HC, WC/HC, ICO, BMI), Glucose and Lipid profile (TC, LDL-C, HDL-C, TG, non-HDL cholesterol, risk ratios), Estimated CVD risk changes (EAS/ESC SCORE Charts), Measures of vascular health (FMD, PWA, PWV, Aix), Liver and renal functionality biomarkers, 24-h urine collection at baseline of treatment phase 1 and endpoint of the final phase will be analysed to account for potential confounding of urinary sodium excretion (intake) As required by the GCPs and GLPs, all the SOPs have already been established and all the personnel to be involved in the study is continuously trained in trials with similar outcomes

ELIGIBILITY:
Inclusion Criteria:

* Primary prevention for cardiovascular diseases
* Systolic blood pressure 130-139 mmHg and/or Diastolic blood pressure 85-89 mmHg
* Estimated cardiovascular risk >5% (Italian Heart Project cards)
* Ability of the volunteer to understand the study finalities and to adhere to the study protocol
* Signed informed consent

Exclusion Criteria:

* Secundary prevention for cardiovascular disease or high risk to develop cardiovascular disease
* Diabetes mellitus
* High level of a single cardiovascular disease risk factor (i.e.: severe hypertension/hypercholesterolemia)
* Chronic renal or liver failure
* Obesity (Body Mass Index>30 kg/m2)
* Coeliac disease or gluten intolerance
* Assumption of antihypertensive drugs at antihypertensive dosage• Each medical or surgery condition potentially making difficult or inconstant the volunteer adhesion to the study protocol

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Office blood pressure modification | 4 weeks
  Systolic, diastolic, pulse, mean arterial pressure, pulse pressure index, mean of 3 consecutive measurement as for the European guidelines on blood pressure measurement suggestion

SECONDARY OUTCOMES:
24-hour blood pressure modification (ABPM) | 4 weeks
  Twenty-four hour ambulatory blood pressure monitoring (ABPM) will be performed using a non-invasive automatic monitor (Space Labs, model 90207). For ABPM, patients will be instructed to act and work as normal between 6:00 AM and 10:00 PM and rest or sleep between 10:00 PM and 6:00 AM. Readings were obtained automatically at 15-min intervals throughout a 24-h study period. Separate averages will be obtained for the 24-h, daytime (6:00 AM-10:00 PM) and night-time (10:00 PM-6:00 AM) values. The accuracy of the automatic blood pressure readings will be checked against manual readings taken using a standard mercury sphygmomanometer, twice for each ABPM. Blood pressure were was measured with the patient sitting, before the beginning of the ABPM, and after a 5-min rest period. The accuracy test will be repeated after the end of each 24-h ABPM.
Cholesterolemia modification | 4 weeks
  12-hour fasting Total, LDL, HDL and non HDL-Cholesterol, evaluated with standardized methods
Flow-mediated vasodilation modification | 4 weeks
  Evaluation of endothelial function by automatic measurement executed with the Vicorder Endopath instrument, already validated in previous publications
Fasting glucose modification | 4 weeks
  12-hour fasting plasma glucose evaluated with standardized methods
Pulse Wave Velocity modification | 4 weeks
  Evaluation of arterial stiffness measured as Pulse Wave Velocity and related parameters by the Vicorder instrument, already validated in previous publications
Triglyceridemia modification | 4 weeks
  12-hour fasting triglyceridemia evaluated by standardized lab methos

OTHER OUTCOMES:
Anthropometric measurement changes | 4 weeks
  Height, weight, body mass index, waist circumference, hip circumference, waist/hip ratio, visceral adiposity index, index of central obesity measured from trained personnel following SOPs
Liver parameters modification | 4 weeks
  12-hour liver transaminases, gamma-glutamyl-transferase, Lipid Accumulation Product, and Hepatic Steatosis Index evaluated with standardized methods
Renal function parameter modification | 4 weeks
  12-hour fasting serum uric acid, creatinine, and estimated glomerular filtration rate (CKD-EPI formula) evaluated with standardized methods

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Borghi, MD, Study Director — University of Bologna
Locations (1):
- S. Orsola-Malpighi University Hospital, Bologna, BO, Italy